CLINICAL TRIAL: NCT05279898
Title: Perioperative Multimodal General AnesTHesia Focusing on Specific CNS Targets in Patients Undergoing carDiac surgERies - the PATHFINDER II Study
Brief Title: Perioperative Multimodal General AnesTHesia Focusing on Specific CNS Targets in Patients Undergoing carDiac surgERies
Acronym: PATHFINDERII
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Balachundhar Subramaniam, Balachundhar Subramaniam MD MPH FASA, Principal Investigator, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2021-P-000889
Record Dates: First submitted 2022-02-14; First posted 2022-03-15 (Actual); Results first posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Postoperative Delirium; Hemodynamic Instability; Pain; Neurocognitive Dysfunction
MeSH Terms: conditions — Emergence Delirium; Pain; Cognition Disorders | interventions — Ropivacaine; Ketamine; Remifentanil; Dexmedetomidine; Rocuronium; Propofol

STUDY DESIGN:
Intervention Model Description: Group 1: Control - receives standard of care anesthesia and blinded EEG and Cerebral Oximetry(CO) monitoring Group 2: Intervention - receives MMGA bundle, guided by EEG monitoring, blinded CO will be passively collected
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Multimodal General Anesthesia (MMGA Bundle) - EEG Guided (Experimental): 1. Routine anesthetic induction
  2. Bilateral Pectoro-interfascial block (PIFB) with 20 mL of 0.2% ropivacaine on both sides of the sternum after anesthetic induction but before surgical incision (total of 40mL)
  3. Ketamine (0.1 to 0.2 mg.kg/hr)
  4. Remifentanil (0.05-0.4 mcg/kg/min)
  5. Dexmedetomidine (0.2-0.5 mcg/kg/hr)
  6. Rocuronium intermittent bolus (TOF)
  7. Propofol infusion (15 to 200 mcg/kg/min)
  Postop
  1. Standard pain management protocol
     * IV Acetaminophen
     * IV Hydromorphone/fentanyl boluses as needed per current practice for rescue analgesia
     * Other oral pain medications as per standard of care (Oxycodone, etc)
  2. Dexmedetomidine infusion (0.4-1.4 mcg/kg/hr) - EEG Guided; Infusion continued till extubation
  3. Propofol infusion may be added/used for sedation based on the treating physician's discretion
  4. PIFB on postoperative day 1 (provided they are extubated/getting ready to be extubated)(for intervention group)
  5. Lidocaine patches
  Interventions: Device: EEG Monitoring; Drug: Ropivacaine; Drug: Ketamine; Drug: Remifentanil; Drug: Dexmedetomidine; Drug: Rocuronium; Drug: Propofol
- Standard of Care/Control (No Intervention): EEG monitoring will be blinded, and not guide anesthesiologists. Patients will receive standard/routine anesthesia practice intraoperatively.
  Postoperative Propofol infusion (15 to 200 mcg/kg/min) ± Sevoflurane
  1. Standard pain management protocol
     * IV Acetaminophen (1 gram) x 4 doses at 6 hour intervals starting from 1 hr after ICU arrival
     * IV Hydromorphone/fentanyl boluses as needed per current practice for rescue analgesia
     * Other oral pain medications as per standard of care (Oxycodone, etc)
  2. Dexmedetomidine infusion (0.4-1.4 mcg/kg/hr) - EEG Guided; Infusion continued till extubation
  3. Propofol infusion may be added/used for sedation based on the treating physician's discretion
  4. Lidocaine patches
  5. Parasternal block (PIFB or Transversus Thoracic Plane Block) on Postoperative day 0 - currently incorporated into standard pain management after surgery based on physician discretion

INTERVENTIONS:
Device: EEG Monitoring — Perioperative monitoring, MMGA guided by EEG for intervention group
  Other Names: Sedline Monitoring
  Arms: Multimodal General Anesthesia (MMGA Bundle) - EEG Guided
Drug: Ropivacaine — Intraoperative bilateral PIFB block with 20 mL of 0.2% Ropivicaine on either side of the sternum after anesthetic induction but before surgical incision (total of 40mL) PIFB on postoperative day 1 (provided they are extubated or getting ready to be extubated) to help with mobilization (for intervention group)
  Arms: Multimodal General Anesthesia (MMGA Bundle) - EEG Guided
Drug: Ketamine — Intraoperative infusion
  Arms: Multimodal General Anesthesia (MMGA Bundle) - EEG Guided
Drug: Remifentanil — Intraoperative infusion
  Arms: Multimodal General Anesthesia (MMGA Bundle) - EEG Guided
Drug: Dexmedetomidine — Intraoperative infusion
  Arms: Multimodal General Anesthesia (MMGA Bundle) - EEG Guided
Drug: Rocuronium — Intraoperative intermittent bolus
  Arms: Multimodal General Anesthesia (MMGA Bundle) - EEG Guided
Drug: Propofol — Intraoperative infusion
  Arms: Multimodal General Anesthesia (MMGA Bundle) - EEG Guided

SUMMARY:
In the PATHFINDER 2 trial, the study investigators will test the intraoperative EEG-guided multimodal general anesthesia (MMGA) management strategy in combination with a postoperative protocolized analgesic approach to:

1. reduce the incidence of perioperative neurocognitive dysfunction in cardiac surgical patients
2. ensure hemodynamic stability and decrease use of vasopressors in the operating rooms
3. reduce pain and opioid consumption postoperatively

DETAILED DESCRIPTION:
The investigators propose to randomize (1:1) 70 patients undergoing cardiac surgery to the perioperative EEG-guided MMGA bundle (described in full below) or standard-of-care management based primarily on the use of sevoflurane for unconsciousness and intermittent doses of fentanyl and hydromorphone for antinociception.

The team will test the intraoperative EEG-guided MMGA management strategy in combination with a postoperative protocolized analgesic approach to reduce the postoperative increase of surgical and delirium markers, reduce intraoperative abnormalities in brain health monitoring, ensure hemodynamic stability and decreased use of vasopressors in the operating rooms and reduce pain and opioid consumption postoperatively. The team will also investigate whether EEG-guided MMGA strategy reduces the incidence of perioperative neurocognitive dysfunction in cardiac surgical patients. This approach will further individualize care and minimize the use of intraoperative vasopressor-inotropic dose, dose of anesthetic medications, and postoperative opioids given to each patient potentially preventing hemodynamic complications and post-operative cognitive dysfunction after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 60 years
* Undergoing any of the following types of surgery with cardiopulmonary bypass limited to coronary artery bypass surgery (CABG), CABG+valve surgeries and isolated valve surgeries.

Exclusion Criteria:

* Preoperative left ventricular ejection fraction (LVEF) <30%
* Emergent surgery
* Non-English speaking
* Cognitive impairment as defined by total MoCA score < 10
* Currently enrolled in another interventional study that could impact the primary outcome, as determined by the PI
* Significant visual impairment
* Chronic opioid use for chronic pain conditions with tolerance (total dose of an opioid at or more than 30 mg morphine equivalent for more than one month within the past year)
* Hypersensitivity to any of the study medications
* Known history of alcohol (> 2 drinks per day) or drug abuse Active (in the past year) history of alcohol abuse (≥5 drinks/day for men or ≥4 drinks/day for women) as determined by reviewing medical record and history given by the patient
* Liver dysfunction (liver enzymes > 4 times the baseline, all patients will have a baseline liver function test evaluation), history and examination suggestive of jaundice.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2023-02-28 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Balachundhar Subramaniam, MD,MPH,FASA, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Background] Brown EN, Lydic R, Schiff ND. General anesthesia, sleep, and coma. N Engl J Med. 2010 Dec 30;363(27):2638-50. doi: 10.1056/NEJMra0808281. No abstract available. PMID 21190458
- [Background] Berger M, Terrando N, Smith SK, Browndyke JN, Newman MF, Mathew JP. Neurocognitive Function after Cardiac Surgery: From Phenotypes to Mechanisms. Anesthesiology. 2018 Oct;129(4):829-851. doi: 10.1097/ALN.0000000000002194. PMID 29621031
- [Background] Brown EN, Pavone KJ, Naranjo M. Multimodal General Anesthesia: Theory and Practice. Anesth Analg. 2018 Nov;127(5):1246-1258. doi: 10.1213/ANE.0000000000003668. PMID 30252709
- [Background] Volkow ND, Collins FS. The Role of Science in Addressing the Opioid Crisis. N Engl J Med. 2017 Jul 27;377(4):391-394. doi: 10.1056/NEJMsr1706626. Epub 2017 May 31. No abstract available. PMID 28564549
- [Background] Mulier J. Opioid free general anesthesia: A paradigm shift? Rev Esp Anestesiol Reanim. 2017 Oct;64(8):427-430. doi: 10.1016/j.redar.2017.03.004. Epub 2017 Apr 18. No abstract available. English, Spanish. PMID 28431750
- [Background] MacKenzie KK, Britt-Spells AM, Sands LP, Leung JM. Processed Electroencephalogram Monitoring and Postoperative Delirium: A Systematic Review and Meta-analysis. Anesthesiology. 2018 Sep;129(3):417-427. doi: 10.1097/ALN.0000000000002323. PMID 29912008
- [Background] Wildes TS, Mickle AM, Ben Abdallah A, Maybrier HR, Oberhaus J, Budelier TP, Kronzer A, McKinnon SL, Park D, Torres BA, Graetz TJ, Emmert DA, Palanca BJ, Goswami S, Jordan K, Lin N, Fritz BA, Stevens TW, Jacobsohn E, Schmitt EM, Inouye SK, Stark S, Lenze EJ, Avidan MS; ENGAGES Research Group. Effect of Electroencephalography-Guided Anesthetic Administration on Postoperative Delirium Among Older Adults Undergoing Major Surgery: The ENGAGES Randomized Clinical Trial. JAMA. 2019 Feb 5;321(5):473-483. doi: 10.1001/jama.2018.22005. PMID 30721296
- [Background] Nicolini F, Agostinelli A, Vezzani A, Manca T, Benassi F, Molardi A, Gherli T. The evolution of cardiovascular surgery in elderly patient: a review of current options and outcomes. Biomed Res Int. 2014;2014:736298. doi: 10.1155/2014/736298. Epub 2014 Apr 10. PMID 24812629
- [Background] Mahanna-Gabrielli E, Schenning KJ, Eriksson LI, Browndyke JN, Wright CB, Culley DJ, Evered L, Scott DA, Wang NY, Brown CH 4th, Oh E, Purdon P, Inouye S, Berger M, Whittington RA, Price CC, Deiner S. State of the clinical science of perioperative brain health: report from the American Society of Anesthesiologists Brain Health Initiative Summit 2018. Br J Anaesth. 2019 Oct;123(4):464-478. doi: 10.1016/j.bja.2019.07.004. Epub 2019 Aug 19. PMID 31439308
- [Background] Maheshwari K, Ahuja S, Khanna AK, Mao G, Perez-Protto S, Farag E, Turan A, Kurz A, Sessler DI. Association Between Perioperative Hypotension and Delirium in Postoperative Critically Ill Patients: A Retrospective Cohort Analysis. Anesth Analg. 2020 Mar;130(3):636-643. doi: 10.1213/ANE.0000000000004517. PMID 31725024
- [Background] Ni K, Cooter M, Gupta DK, Thomas J, Hopkins TJ, Miller TE, James ML, Kertai MD, Berger M. Paradox of age: older patients receive higher age-adjusted minimum alveolar concentration fractions of volatile anaesthetics yet display higher bispectral index values. Br J Anaesth. 2019 Sep;123(3):288-297. doi: 10.1016/j.bja.2019.05.040. Epub 2019 Jul 3. PMID 31279479
- [Background] Hesse S, Kreuzer M, Hight D, Gaskell A, Devari P, Singh D, Taylor NB, Whalin MK, Lee S, Sleigh JW, Garcia PS. Association of electroencephalogram trajectories during emergence from anaesthesia with delirium in the postanaesthesia care unit: an early sign of postoperative complications. Br J Anaesth. 2019 May;122(5):622-634. doi: 10.1016/j.bja.2018.09.016. Epub 2018 Oct 25. PMID 30915984
- [Background] Shanker A, Abel JH, Narayanan S, Mathur P, Work E, Schamberg G, Sharkey A, Bose R, Rangasamy V, Senthilnathan V, Brown EN, Subramaniam B. Perioperative Multimodal General Anesthesia Focusing on Specific CNS Targets in Patients Undergoing Cardiac Surgeries: The Pathfinder Feasibility Trial. Front Med (Lausanne). 2021 Oct 14;8:719512. doi: 10.3389/fmed.2021.719512. eCollection 2021. PMID 34722563

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants undergoing elective cardiac surgery were recruited from a tertiary academic hospital between February 28, 2023, and December 31, 2024, for a randomized trial comparing EEG-guided multimodal general anesthesia with standard care. Recruitment occurred in preoperative clinics, inpatient wards, and surgical units.
Pre-assignment Details: There were no washout, run-in, or lead-in phases. All enrolled participants were randomized in a 1:1 ratio to either the EEG-guided multimodal general anesthesia (MMGA) group or the standard care group without pre-assignment exclusions.
Period: Overall Study
Arm/Group | Multimodal General Anesthesia (MMGA Bundle) - EEG Guided | Standard of Care/Control
Started | 35 | 35
Surgery | 33 | 34
1 month Follow-up | 19 | 23
6 month Follow-up | 18 | 21
Completed (For Primary Outcome) | 33 | 34
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Physician Decision | 1 | 1

BASELINE CHARACTERISTICS:
Population: One participant's baseline information is missing in the intervention group, and one participant's ethnicity data is missing in the control group
Groups:
- Total: Total of all reporting groups
Arm/Group | Multimodal General Anesthesia (MMGA Bundle) - EEG Guided | Standard of Care/Control | Total
Number analyzed (Participants) | 34 | 35 | 69
Age, Continuous [Mean (Standard Deviation); unit: years] — Baseline measure values were compared between groups using the Wilcoxon rank-sum exact test, a nonparametric statistical test that assesses whether two independent samples come from the same distribution. This method does not assume normality and is appropriate for ordinal or continuous data that may not follow a normal distribution Population: One participant's baseline information is missing in the intervention group
  years | 70 (6) | 71 (7) | 70.507 (6.50)
Sex: Female, Male [Count of Participants; unit: Participants] — Baseline sex distribution was compared between groups using Fisher's exact test, a statistical method for assessing the association between categorical variables, especially appropriate for small sample sizes Population: One participant's baseline information is missing in the intervention group
  Participants
    Female | 5 | 8 | 13
    Male | 29 | 27 | 56
Race (NIH/OMB) [Count of Participants; unit: Participants] — Baseline Race was compared between groups using Fisher's exact test, a statistical method for assessing the association between categorical variables, especially appropriate for small sample sizes Population: One participant's baseline information is missing in the intervention group
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 2 | 1 | 3
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 2 | 1 | 3
    White | 30 | 33 | 63
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Baseline Ethnicity was compared between groups using Fisher's exact test, a statistical method for assessing the association between categorical variables, especially appropriate for small sample sizes Population: One participant's baseline information is missing in the intervention group, and one participant's ethnicity data is missing in the control group
  Participants
    number analyzed (Participants) | 34 | 34 | 68
    Hispanic or Latino | 1 | 0 | 1
    Not Hispanic or Latino | 33 | 34 | 67
    Unknown or Not Reported | 0 | 0 | 0
Baseline plasma IL-6 and NFL Levels [Mean (Standard Deviation); unit: pg/mL] — Plasma interleukin-6 (IL-6) and Neurofilament Light (NFL) levels will be measured at baseline Population: The number of participants analyzed at each time point differs from the number originally assigned due to missing or inadequate biospecimen samples for IL-6 and NFL measurements at baseline. Participants without valid samples at a given time point were excluded from that specific analysis.
  pg/mL
    IL-6 - Baseline: number analyzed (Participants) | 34 | 32 | 66
    IL-6 - Baseline | 15 (28.5) | 29.5 (79.9) | 22.03 (59.15)
    NFL Baseline: number analyzed (Participants) | 34 | 32 | 66
    NFL Baseline | 40.9 (37.1) | 28.6 (37.4) | 34.93 (37.48)

OUTCOME MEASURES:

1. Primary Outcome: Increase in Plasma IL-6 Levels
Description: Plasma interleukin-6 (IL-6) levels will be measured at baseline, postoperative day 1, and postoperative day 2. The change in IL-6 concentration from baseline to each postoperative time point will be calculated and compared between the study groups.
Time Frame: Baseline, postoperative day 1, and postoperative day 2
Population: The number of participants analyzed at each time point differs from the number originally assigned due to missing or inadequate biospecimen samples for IL-6 and NFL measurements at baseline and postoperative days 1 and 2. Participants without valid samples at a given time point were excluded from that specific analysis.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Multimodal General Anesthesia (MMGA Bundle) - EEG Guided | Standard of Care/Control
Number analyzed (Participants) | 34 | 32
pg/mL
  IL-6 - Baseline | 15 (28.5) | 29.5 (79.9)
  Il-6 - POD1: number analyzed (Participants) | 33 | 32
  Il-6 - POD1 | 80.5 (65.4) | 97.7 (93.5)
  IL-6 - POD2: number analyzed (Participants) | 31 | 29
  IL-6 - POD2 | 115.7 (64.1) | 164 (108.7)

2. Primary Outcome: Increase in Plasma Neurofilament Light Levels
Description: Plasma neurofilament light (NfL) levels will be measured at baseline, postoperative day 1, and postoperative day 2. The change in NfL concentration from baseline to each postoperative time point will be calculated and compared between the study groups.
Time Frame: Baseline, postoperative day 1, and postoperative day 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Multimodal General Anesthesia (MMGA Bundle) - EEG Guided | Standard of Care/Control
Number analyzed (Participants) | 34 | 32
pg/mL
  NFL - Baseline | 40.9 (37.1) | 28.6 (37.4)
  NFL - POD1: number analyzed (Participants) | 33 | 32
  NFL - POD1 | 37.4 (39.5) | 25.8 (23.2)
  NFL - POD2: number analyzed (Participants) | 31 | 29
  NFL - POD2 | 56.8 (49.3) | 52.8 (46.5)

3. Secondary Outcome: Opioid Consumption
Description: Total opioid consumption during the first 48 postoperative hours will be calculated by summing all opioid doses administered in any route and converting to intravenous morphine milligram equivalents (MME) for standardization. The cumulative 48-hour opioid dose will be compared between groups.
Time Frame: From end of surgery to 48 hours postoperatively
Population: 2 subjects in intervention group and 1 subject in control group withdrew from study after the consent before the start of study procedure
Measure: Mean (Standard Deviation); unit: Morphine Milligram Equivalents (MME)
Arm/Group | Multimodal General Anesthesia (MMGA Bundle) - EEG Guided | Standard of Care/Control
Number analyzed (Participants) | 33 | 34
Morphine Milligram Equivalents (MME) | 132.42 (77.05) | 126.93 (58.12)

4. Secondary Outcome: Pain Scores
Description: Postoperative pain intensity will be assessed using the Numeric Rating Scale (NRS), a validated 11-point scale that measures patient-reported pain intensity from 0 to 10, where 0 indicates no pain and 10 indicates the worst possible pain. Scores will be obtained by nursing staff every 4-8 hours from electronic medical records, and the average 48-hour postoperative pain score will be compared between groups.
Time Frame: From end of surgery to 48 hours postoperatively
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Multimodal General Anesthesia (MMGA Bundle) - EEG Guided | Standard of Care/Control
Number analyzed (Participants) | 33 | 34
Scores on a scale | 4.33 (1.56) | 4.72 (1.69)

5. Secondary Outcome: Burst Suppression
Description: Duration of burst suppression was extracted and quantified from the intraoperative EEG record and compared between the MMGA and control groups.
Time Frame: intraoperative period, from anesthetic induction until the end of surgery
Population: 5 subjects from the intervention group and 4 subjects in control group are removed from analysis due to artifacts in EEG data
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Multimodal General Anesthesia (MMGA Bundle) - EEG Guided | Standard of Care/Control
Number analyzed (Participants) | 28 | 30
minutes | 4.83 (3.47) | 1.68 (2.2)

6. Secondary Outcome: Postoperative Delirium
Description: Incidence of Postoperative Delirium (POD) will be compared between both groups: POD will be diagnosed by our trained research members based on the Confusion Assessment Method (CAM) algorithm postoperatively until discharge.
Time Frame: From postoperative day 1 until hospital discharge, an average of 4 days
Measure: Number; unit: Participants with delirium
Arm/Group | Multimodal General Anesthesia (MMGA Bundle) - EEG Guided | Standard of Care/Control
Number analyzed (Participants) | 33 | 33
Participants with delirium | 8 (2.6) | 9 (2.78)

7. Secondary Outcome: Cognitive Function
Description: Postoperative cognitive function will be assessed at 1 and 6 months after surgery using the telephone version of the Montreal Cognitive Assessment (t-MoCA). The t-MoCA has a total score range of 0 to 22, where higher scores indicate better cognitive function.
Time Frame: Patients will be assessed for cognitive function at 1 month and 6 months following the date of surgery
Population: Lost to follow-up
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Multimodal General Anesthesia (MMGA Bundle) - EEG Guided | Standard of Care/Control
Number analyzed (Participants) | 20 | 25
scores on a scale
  1 month follow-up | 18.421 (2.631) | 18.174 (2.855)
  6 month follow-up | 18.100 (2.075) | 18.960 (1.767)

8. Secondary Outcome: Hemodynamic Stability - Total Vasopressor Dose
Description: Metrics of total vasopressor dose in norepinephrine equivalents (mcg/kg/min) will be collected from the intra-operative record and medical records to be quantified and compared.
Time Frame: Intraoperative period, from induction of anesthesia until transfer from the operating room
Population: 3 subjects change of consent status before surgery
Measure: Mean (Standard Deviation); unit: norepinephrine equivalents (mcg/kg/min)
Arm/Group | Multimodal General Anesthesia (MMGA Bundle) - EEG Guided | Standard of Care/Control
Number analyzed (Participants) | 33 | 34
norepinephrine equivalents (mcg/kg/min) | 1109.425 (2311.095) | 2358.042 (4543.262)

ADVERSE EVENTS:
Time Frame: From the day of surgery until postoperative day 4
Description: Adverse events were defined and collected per institutional CCI policy, which may differ slightly from ClinicalTrials.gov definitions. Events were recorded daily during hospitalization for up to four postoperative days, regardless of relatedness, and included both serious and non-serious events. Structured assessments captured clinical events such as arrhythmias, hypotension, infection, hematoma, and local anesthetic systemic toxicity. Analyses included all participants who received the assigned
Arm/Group | Multimodal General Anesthesia (MMGA Bundle) - EEG Guided | Standard of Care/Control
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/34
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/34
Other Adverse Events (participants affected / at risk) | 0/33 | 0/34

LIMITATIONS AND CAVEATS:
This single-center trial enrolled a small sample and was not powered for clinical outcomes such as delirium. Some biomarker and EEG data were missing or artifact-limited, and anesthesia depth may have differed between groups. These factors may limit generalizability and interpretation of results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-07-05): https://cdn.clinicaltrials.gov/large-docs/98/NCT05279898/Prot_SAP_000.pdf